CLINICAL TRIAL: NCT05384652
Title: Simultaneous Quantification of Liver Fat Content, Fatty Acid Composition, and Fibrosis Using Non-invasive Breath-hold Quantitative Spin-lock MRI for Assessment of Non-Alcoholic Steatohepatitis
Brief Title: Simultaneous Quantification of Liver Fat Content, Fatty Acid Composition, and Fibrosis Using Spin-lock MRI for Steatohepatitis Assessment
Status: Not yet recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chen Weitian, Associate Professor, Chinese University of Hong Kong
Other Study IDs: 2022.021
Record Dates: First submitted 2022-05-17; First posted 2022-05-20 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Non-alcoholic Fatty Liver Disease (NAFLD); Non-alcoholic Steatohepatitis (NASH)
Keywords: chronic liver diseases; liver fibrosis; fatty acid; spin-lock MRI; non-invasive imaging
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- subjects with NASH
- subjects with simple steatosis
- healthy subjects

SUMMARY:
Non-alcoholic fatty liver disease is a major health problem worldwide. It includes simple steatosis and NASH which has inflammation in the liver, with or without fibrosis. Fat content, fibrosis, and inflammation are three important components to evaluate NASH. Liver biopsy is the current gold standard for the diagnosis of NASH. Liver biopsy; however, is invasive. The existing non-invasive methods still have significant limitations to assess NASH. It was reported that quantification of fatty acid composition is feasible for evaluation of metabolic disorders and inflammatory conditions. However, this measurement cannot be used to evaluate fibrosis. Liver fibrosis is characterized by excessive deposition of collagen-rich connective tissues in the liver, which can be quantified by macromolecular proton fraction (MPF), an MRI parameter reflecting the macromolecular level in tissues. Although it has the potential to directly quantify fibrotic tissue, the effect of inflammation on MPF measurement was not well studied. In summary, NASH assessment using non-invasive imaging methods remains challenging. Based on our previous work of MPF imaging with spin-lock (MPF-SL) and chemical-shift encoding-based water-fat imaging in spin-lock MRI, the investigators will develop a fast acquisition technology to collect data for simultaneous quantification of liver fat content, fatty acid composition, and fibrosis within a single breath-hold less than 14 seconds. Our method does not require extra hardware and does not need to inject a contrast agent. The investigators will evaluate the repeatability and reproducibility of the proposed method on volunteers. To evaluate its clinical value, the investigators will recruit 120 subjects (60 with simple steatosis and 60 with NASH) in this study. The investigators will use histology analysis as the gold standard and evaluate the diagnostic value of our proposed method for detecting NASH. This project will provide a non-invasive diagnostic technology for the assessment of NASH. The proposed MRI technology also has the potential to be applied for other clinical purposes.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 65 years of age.
* Non-alcoholic fatty liver disease (NAFLD) patients at stage of either Non-alcoholic steatohepatitis (NASH) or simple steatosis
* NAFLD patients scheduled to undergo liver biopsy.
* No abnormal lesions detected at baseline MRI exam for healthy volunteers.

Exclusion Criteria:

* Evidence of hepatocarcinoma (HCC) or any other types of neoplasm.
* Patients who had undergone liver transplantation.
* Any contraindications to either liver biopsy or MRI scan.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: subjects with NASH or with simple steatosis
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
To simultaneously quantify macromolecular proton fraction, proton density fat fraction, and fatty acid composition in liver tissues | one year
  The MRI technology developed can serve as a non-invasive, fast, and robust imaging tool to simultaneously quantify macromolecular proton fraction, proton density fat fraction, and fatty acid composition in liver tissues.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Prince of Wale Hospital, Hong Kong, Shatin, Hong Kong